CLINICAL TRIAL: NCT00907166
Title: A Phase I/II Open-Label Dose-Escalation Clinical Trial of CPI-613 in Combination With Gemcitabine in Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Suspended trial was not restarted.
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-CPI-613-004
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Cancer; Pancreatic Cancer; Pancreatic Carcinoma
Keywords: Cornerstone Pharmaceuticals, Inc.; CPI-613; Altered Energy Metabolism Directed Compound; Phase I; Phase II; Cancer; Carcinoma of the Pancreas; Pancreatic Cancer; Pancreatic Carcinoma
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms | interventions — devimistat; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase I, Arm A (Experimental): CPI-613 + Gemcitabine
  Interventions: Drug: CPI-613; Drug: Gemcitabine
- Phase II, Arm A (Experimental): CPI-613 + Gemcitabine
  Interventions: Drug: CPI-613; Drug: Gemcitabine
- Phase II, Arm B (Active Comparator): Gemcitabine
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: CPI-613 — IV infusion of CPI-613 given on Days 1,4, 8, 11, 15, 18, of 28 day cycle in cancer patients.
  Arms: Phase I, Arm A
Drug: CPI-613 — IV infusion of CPI-613 given on Days 1, 4, 8, 11, 15, 18, of 28 day cycle in patients with pancreatic carcinoma.
  Arms: Phase II, Arm A
Drug: Gemcitabine — IV infusion of 1000 mg/m^2 of Gemcitabine given on Days 1, 8, and 15 of a 28 day cycle in patients with pancreatic carcinoma.
  Arms: Phase II, Arm B
Drug: Gemcitabine — IV infusion of 1000 mg/m^2 of Gemcitabine given on Days 1, 8, and 15 of a 28 day cycle in cancer patients.
  Arms: Phase I, Arm A
Drug: Gemcitabine — IV infusion of 1000 mg/m^2 of Gemcitabine given on Days 1, 8, and 15 of a 28 day cycle in patients with pancreatic carcinoma.
  Arms: Phase II, Arm A

SUMMARY:
The objectives of this study are:

* To determine the safety and MTD of CPI-613, when used in combination with Gemcitabine, in cancer patients.
* To compare the safety and efficacy of CPI-613/Gemcitabine combination vs. Gemcitabine alone in patients with carcinoma of the pancreas.

DETAILED DESCRIPTION:
CPI-613, the investigational drug, is a novel anti-tumor compound believed to operate via a novel mechanism of action that does not belong to any existing pharmacological class of anticancer agents currently being used in the clinics. Specifically, CPI-613 is Cornerstone Pharmaceutical Inc.'s lead drug from its Altered Energy Metabolism-Directed (AEMD) technology platform. It is selective against tumor cells (but not normal cells)according to preclinical studies.

ELIGIBILITY:
Inclusion Criteria:

* For Stages 1 and 2 of the study, histologically documented unresectable primary or metastatic carcinoma of the pancreas, Stage II-IV, diagnosed within the past 8 weeks, intended to be treated with Gemcitabine as a single agent at 1000 mg/m^2 once weekly for 3 weeks repeating the cycle every 4 weeks. For Stage 1 but not Stage 2 of the study, patients also include those with histologically documented unresectable primary or metastatic carcinoma other than pancreatic carcinoma (e.g., bladder cancer, NSCLC, and biliary tract cancer) who are intended to be treated with Gemcitabine as a single agent at 1000 mg/m^2 once weekly for 3 weeks repeating the cycle every 4 weeks, regardless if Gemcitabine is used as second, third or fourth line treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status being 0-2.
* Expected survival >2 months.
* 18-70 years of age of both genders
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
* No radiotherapy, treatment with cytotoxic agents or chemotherapeutic agents (except CPI-613), or treatment with biologic agents within the 2 weeks prior to treatment with CPI-613. At least 2 weeks must have elapsed from any prior surgery or hormonal therapy. Patients must have fully recovered from the acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤Grade 1 are eligible, but must be documented as such.
* Laboratory values ≤2 weeks must be:

  * Adequate hematologic (white blood cell [WBC] ≥3500 cells/mm^3 or ≥3.5 bil/L; platelet count ≥150,000 cells/mm^3 or ≥150 bil/L; absolute neutrophil count [ANC] ≥1500 cells/mm3 or ≥1.5 bil/L; and hemoglobin ≥9 g/dL or ≥90 g/L).
  * Adequate hepatic function (aspartate aminotransferase [AST/SGOT] ≤3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] ≤3x UNL (≤5x UNL if liver metastases present), bilirubin ≤3x UNL).
  * Adequate renal function (serum creatinine ≤2.0 mg/dL or 177 µmol/L).
  * Adequate coagulation (International Normalized Ratio or INR must be≤1.5)
* No evidence of active infection and no serious infection within the past month.
* Mentally competent, ability to understand and willingness to sign the informed consent form.

Exclusion Criteria:

* Prior therapy with Gemcitabine
* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity.
* Patients with active central nervous system (CNS) or epidural tumor.
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease).
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown).
* Lactating females.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Life expectancy less than 2 months.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.
* Unwilling or unable to follow protocol requirements.
* Dyspnea with minimal to moderate exertion. Patients with large pleural, pericardial, or peritoneal effusions.
* Active heart disease including myocardial infarction within previous 6 months, symptomatic coronary artery disease, arrhythmias requiring medication, or symptomatic congestive heart failure.
* Albumin <2.5 g/dL or <25 g/L.
* Evidence of active infection, or serious infection within the past month.
* Patients with known HIV infection.
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 4 weeks prior to initiation of CPI-613 treatment.
* Patients who have received immunotherapy of any type within the past 4 weeks prior to initiation of CPI-613 treatment.
* Requirement for immediate palliative treatment of any kind including surgery.
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months.
* A marked baseline prolongation of QT/QTc interval (e.g., repeated exhibition of a QTc interval >470 ms.)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Prior illicit drug addiction.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and MTD of CPI-613, when used in combination with Gemcitabine, in cancer patients. | 1 Year

SECONDARY OUTCOMES:
To compare the safety and efficacy of CPI-613 Gemcitabine combination vs. Gemcitabine alone in patients with carcinoma of the pancreas. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Avi Retter, M.D., Principal Investigator — Eastchester Center for Cancer Care; Neil Senzer, M.D., Principal Investigator — Mary Crowley Cancer Research Centers
Locations (2):
- United States (2):
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Mary Crowley Cancer Research Centers, Dallas, Texas